CLINICAL TRIAL: NCT00672217
Title: Cognitive-Behavioral Therapy for Chronic Insomnia After Breast Cancer Treatment
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Denver Health Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07-0924; 5K23NR010587 (NIH)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer survivors, insomnia, quality of life
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Placebo Therapy (Placebo Comparator): Behavioral Placebo Treatment
  Interventions: Behavioral: Behavioral Placebo Treatment
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy for Insomnia (CBTI)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI) — Six 15-30 minute in-person or phone sessions that incorporate cognitive, behavioral and psycho-educational techniques focused on modifying the perpetuating factors that maintain insomnia.
  Arms: Cognitive Behavioral Therapy
Behavioral: Behavioral Placebo Treatment — Six 15-30 minute in-person or phone sessions that begin with a review of the sleep diary, a general discussion of treatment progress and tabulation of sleep parameters.
  Arms: Behavioral Placebo Therapy

SUMMARY:
The primary goal of the proposed study is to examine a cognitive behavioral intervention for insomnia (CBTI) in women after breast cancer treatment. Chronic Insomnia is a highly prevalent and distressing symptom in cancer patients. CBTI is considered the treatment of choice for chronic primary insomnia. Few studies have been conducted in cancer survivors to evaluate the effect of CBTI on sleep and clinically relevant outcomes.

DETAILED DESCRIPTION:
The overall goals of this study are to: 1) test standard 4-component CBTI in patients with breast cancer post-treatment, 2) gather data on the feasibility of the methods, and 3) determine effects of the intervention on quality of life (QOL) and daily functioning. Sixty women after completion of primary breast cancer treatment, 21-65 years of age, who meet the criteria for chronic insomnia will be recruited from two Western U.S. Cancer Centers. Participants will be randomized to one of two treatment conditions (CBTI or behavioral placebo treatment). Both groups will receive six in-office and phone sessions. The control group will receive the same amount of individualized attention. Sleep efficiency and component measures (e.g., sleep onset latency, minutes awake after sleep onset) and quality of life and component measures of daily functioning will be assess pre and post-intervention, and at 3- and 6-month follow up visits. It is hypothesized that women receiving CBTI treatment will demonstrate greater increase in sleep efficiency (time in bed compared with time asleep) and will self-report greater improvements in QOL and daily functioning compared to those receiving a behavioral placebo treatment at the conclusion of the intervention and at 3- to 6-month follow-ups. Established instruments include the Insomnia Severity Index, Morin Sleep Diary, Dysfunctional Beliefs and Attitudes about Sleep-16, European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30, Attentional Function Index, Revised Piper Fatigue Scale, and Hospital Anxiety and Depression Scale. Subjective data will be corroborated with actigraphy. Results may inform development of clinical guidelines for insomnia management after cancer treatment. The proposed study associated with this K23 award relates to the Health People 2010 goal of improving quality of life of individuals of all ages, and the cancer focus area goal of reducing illness and disability caused by cancer.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years of age inclusive
* 1-36 months after radiation or chemotherapy for non-metastatic breast cancer and on a stable dose of anti-estrogen agent and medications for hot flashes
* Meets diagnostic criteria for chronic, secondary insomnia
* Speak and write English

Exclusion Criteria:

* Presence of a serious unstable physical illness other than cancer
* Presence of dementia, major depression, psychosis or other serious psychiatric disorder
* Presence of a sleep disorder other than insomnia
* Unstable doses of psychotropic medications (excluding hypnotics), opioids, anit-endocrine medications, or use of high dose steroids
* Current evening/night shift employment

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
sleep efficiency | baseline, pre and post intervention, 3-months, 6-months

SECONDARY OUTCOMES:
sleep latency, total sleep time, quality of life, fatigue | baseline, pre and post intervention, 3-months, 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Ellyn E Matthews, PhD,RN,AOCN, Principal Investigator — University of Colorado, Denver College of Nursing
Locations (1):
- University of Colorado, College of Nursing, Aurora, Colorado, United States

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811